CLINICAL TRIAL: NCT00156013
Title: A Phase I/II Open-label Study of Clofarabine in Patients With Relapsed or Refractory Diffuse Large Cell B-Cell NHL
Brief Title: Clofarabine for Relapsed or Refractory T-Cell or B-Cell Non-Hodgkin Lymphoma (NHL)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Oncology Specialists, S.C. (Other)
Collaborators: Genzyme, a Sanofi Company (Industry)
Responsible Party: Principal Investigator, Dr. Sigrun Hallmeyer, Principal Investigator, Oncology Specialists, S.C.
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1066306 (0408); NCT00305721 (obsolete NCT alias)
Record Dates: First submitted 2005-09-08; First posted 2005-09-12 (Estimated); Results first posted 2012-07-09 (Estimated); Last update posted 2017-11-29 (Actual); Status verified 2017-10

CONDITIONS: Lymphoma, B-Cell; Lymphoma, Non-Hodgkin
Keywords: B-Cell NHL
MeSH Terms: conditions — Lymphoma, B-Cell; Lymphoma, Non-Hodgkin | interventions — Clofarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): Clofarabine 4 mg/m^2 days 1-5 of every cycle for a maximum of 6 cycles.
  Interventions: Drug: CLOFARABINE

INTERVENTIONS:
Drug: CLOFARABINE — 4 mg/m^2 days 1-5 of every cycle for a maximum of 6 cycles
  Other Names: Clolar®

SUMMARY:
This research is being done to develop new treatment for non-hodgkin's lymphoma in subjects whose cancer has returned or resisted treatment with chemotherapy. The investigational drug clofarabine is being used in this study. An investigational drug is one that has not been approved by the United States Food and Drug Administration (FDA).

DETAILED DESCRIPTION:
The safety profile of clofarabine appears acceptable within the target populations studied to date in the clinical studies, with numerous responses observed in heavily pre-treated patients with relapsed/refractory ALL or AML. Dose escalation of clofarabine in patients with solid tumors and lymphoproliferative disorders has been limited because grade 3 and 4 myelosuppression was considered acceptable in patients with acute leukemia, provided that hematologic recovery occurred within 6 weeks of therapy , and dose escalation has proceeded as high as 40 mg/m2 in this patient population. Furthermore, no responses were observed in a recent trial in which patients with relapsed CLL were treated with clofarabine 2 mg/m2, an indolent B-cell lymphoproliferative disorder indicating that low doses are likely to be ineffective in patients with aggressive NHL. (Personal Communication with ILEX Products, INC.)

This Phase I/II study will evaluate escalating doses of clofarabine in patients with relapsed and refractory diffuse large cell B-cell NHL starting at a dose of 4 mg/m2/day for 5 consecutive days and repeated every 28 days for a maximum of 6 cycles. This dosing regimen should be evaluated in this patient population because there is no standard therapy at relapse and grade 3 and 4 myelosuppression is frequently observed with traditional NHL salvage. Additionally, patients will receive granulocyte colony stimulating factors at the discretion of the investigator. Antifungal and antibacterial prophylaxis will be administered to minimize the risk of infection.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients who are at least 18 years old with histology confirmed diffuse large cell B-cell NHL who have failed prior systemic chemotherapy with or without monoclonal antibody-based therapies.
* Measurable disease determined by Ct or PET scans or bone marrow involvement, defined as lesions that can be accurately measured in two dimensions by CT or PET scan with the longest diameter accurately as greater than or equal to 1.0 cm or palpable lesions with both diameters greater than or equal to 2.0 cm. PET scan measurable disease is defined based on SUV value as determined by nuclear medicine evaluation.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0,1,or 2.
* Life expectancy greater than 12 weeks.
* Laboratory values obtained less than or equal to 14 days prior to registration:

  * Absolute neutrophil count (ANC) greater than or equal to 1500.
  * White blood cell (WBC) count greater than 3.0.
  * Platelets greater than or equal to 100.
  * Hemoglobin (HG) greater than 9.0 g/dL.
  * Total bilirubin less than or equal to 2.0 mg/dL.
  * Aspartate transaminase (AST)/alanine transaminase (ALT) less than or equal to 3 times the upper limit of normal (ULN). Higher values are acceptable if it is deemed that they are related to liver involvement with NHL.
  * Serum creatinine less than or equal to 2.0 mg/dL.
* Cardiac function on pretreatment MUGA scan or echocardiogram that is considered normal by institutional standards.
* Capable of understanding the investigational nature, potential risks and benefits of the study, and able to provide valid informed consent.
* Female patients of childbearing potential must have a negative serum pregnancy test within 2 weeks prior to enrollment.
* Male and female patients must use an effective contraceptive method during the study and for a minium of 6 months after study treatment.

Exclusion Criteria:

* Previously untreated NHL.
* Received previous treatment with clofarabine.
* History of T-cell lymphoma.
* Bulky disease (ie, any single mass greater than 10 cm or circulating malignant cells greater than or equal to 24,000 cells/ul.
* Patients with known AIDS-related or HIV-positive lymphoma.
* Autologous bone marrow or stem cell transplant within 3 months of study entry.
* History of allogeneic bone marrow transplant or organ transplant.
* Prior radiotherapy to the only site of measurable disease.
* Any medical condition that requires chronic use of oral high-dose corticosteroids. ( in excess of 1 mg/kg/day).
* Autoimmune thrombocytopenia.
* Use if investigational agents within 30 days or any anticancer therapy within 3 weeks before study entry. The patient must have recovered from all acute toxicities from any previous therapy.
* Patients with an active, uncontrolled systemic infection considered to be opportunistic, life threatening, or clinically significant at the time of treatment or with a known or suspected fungal infection (ie, patients of parenteral antifungal therapy).
* HIV-positive status.
* Active secondary malignancy.
* Pregnant or lactating patients.
* Any significant concurrent disease, illness , or psychiatric disorder that would compromise patient safety or compliance, interfere with consent, study participation, follow-up, or interpretation of study results.
* Patients with active or untreated central nervous lymphoma (CNS) lymphoma.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2005-09; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chadi Nabhan, MD, Principal Investigator — Oncology Specialists,SC
Locations (1):
- Oncology Specialists, SC, Park Ridge, Illinois, United States

REFERENCES:
- [Derived] Nabhan C, Davis N, Bitran JD, Galvez A, Fried W, Tolzien K, Foss S, Dewey WM, Venugopal P. Efficacy and safety of clofarabine in relapsed and/or refractory non-Hodgkin lymphoma, including rituximab-refractory patients. Cancer. 2011 Apr 1;117(7):1490-7. doi: 10.1002/cncr.25603. Epub 2010 Nov 8. PMID 21425150

RESULTS

PARTICIPANT FLOW:
Groups:
- Clofarabine: Clofarabine 4 mg/m^2 days 1-5 of every cycle for a maximum of 6 cycles.
Period: Overall Study
Arm/Group | Clofarabine
Started | 33
Completed | 31
Not Completed | 2

BASELINE CHARACTERISTICS:
Arm/Group | Clofarabine
Number analyzed (Participants) | 33
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 13
  >=65 years | 20
Age, Continuous [Mean (Full Range); unit: years] | 69 [27 to 85]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19
  Male | 14
Region of Enrollment [Number; unit: participants]
  United States | 33

OUTCOME MEASURES:

1. Primary Outcome: Phase I Maximum Tolerated Dose
Description: Maximum Tolerated Dose for Clofarabine. Cohorts of 3 patients each will receive doses of clofarabine increased in increments as follows: 4, 6, 8, 10, 12,…etc mg/m2/day for 5 days. The dose level immediately below the MTD will be used to treat patients in the Phase II part of the study. Starting dose of 4 mg/m2.
Time Frame: days 1 -28, maximum 6 cycles
Population: Per protocol guidelines for accrual to the cohorts.
Measure: Number; unit: mg/m^2
Groups:
- Clofarabine: During the Phase I part of the study, the starting dose of clofarabine will be 4 mg/m2 administered by IVI over 1 hour for 5 consecutive days and repeated every 28 days until disease progression is observed or for a maximum of 6 cycles. Cohorts of 3 patients each will receive doses of clofarabine increased in increments of 2mg/m2. The MTD was 6mg/m2. The dose level immediately below the MTD (4mg/m2) will be used to treat patients in the Phase II part of the study.
Arm/Group | Clofarabine
Number analyzed (Participants) | 33
mg/m^2 | 6

2. Primary Outcome: Phase II Overall Response
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.
Time Frame: 5 years
Measure: Count of Participants; unit: Participants
Groups:
- Open Label Trial of Clofarabine in Relapsed or Refractory NHL: Clofarabine 4 mg/m^2 days 1-5 of every cycle for a maximum of 6 cycles.
  CLOFARABINE: 4 mg/m^2 days 1-5 of every cycle for a maximum of 6 cycles
Arm/Group | Open Label Trial of Clofarabine in Relapsed or Refractory NHL
Number analyzed (Participants) | 33
Participants
  patients achieving a complete response | 7
  patients achieving a partial response | 6
  Patients not achieving a response | 20

3. Secondary Outcome: Toxicity
Description: Number of Participants with Toxicity
Time Frame: 5 years
Measure: Count of Participants; unit: Participants
Groups:
- Toxicity: Myelosuppresion
Arm/Group | Toxicity
Number analyzed (Participants) | 33
Participants
  grade 3 or higher neutropenia or thrombocytopenia | 20
  neutropenia or thrombocytopenia less than grade 2 | 13

ADVERSE EVENTS:
Arm/Group | Clofarabine
Serious Adverse Events (participants affected / at risk) | 21/33
Other Adverse Events (participants affected / at risk) | 33/33
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Clofarabine (N=33)
Anemia (Blood and lymphatic system disorders) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 2 (2)
bilateral lower extremity celluiltis (Infections and infestations) | 1 (1)
arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1)
fever of unknown origin (Infections and infestations) | 1 (1)
hyperglycemia (Endocrine disorders) | 1 (1)
hypokalemia (Blood and lymphatic system disorders) | 1 (1)
mental status changes (Psychiatric disorders) | 1 (1)
neutropenic fever (Infections and infestations) | 6 (6)
pancytopenia (Blood and lymphatic system disorders) | 3 (3)
pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 1 (1)
lower back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
renal failure (Renal and urinary disorders) | 1 (1)
renal insufficiency (Renal and urinary disorders) | 1 (1)
seizure (Nervous system disorders) | 1 (1)
syncope (Cardiac disorders) | 1 (1)
thrombocytopenia (Blood and lymphatic system disorders) | 2 (2)
tumor lysis syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
abdominal pain (Musculoskeletal and connective tissue disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Clofarabine (N=33)
abdominal bloating (Musculoskeletal and connective tissue disorders) | 1 (1)
abdominal girth (Musculoskeletal and connective tissue disorders) | 1 (1)
abdominal pain (Musculoskeletal and connective tissue disorders) | 2 (2)
acute renal failure (Renal and urinary disorders) | 1 (1)
Alk Phos (Blood and lymphatic system disorders) | 6 (6)
alopecia (General disorders) | 3 (3)
anemia (Blood and lymphatic system disorders) | 27 (27)
anion gap acidosis (General disorders) | 1 (1)
angina (Cardiac disorders) | 1 (1)
ankle pain (Musculoskeletal and connective tissue disorders) | 1 (1)
anorexia (General disorders) | 2 (2)
anxiety (Psychiatric disorders) | 1 (1)
arm swelling (General disorders) | 1 (1)
back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
bacteremia (Infections and infestations) | 1 (1)
bilateral leg cramping and hand cramping (Musculoskeletal and connective tissue disorders) | 2 (2)
bilateral lower extremity erythema & swelling (Blood and lymphatic system disorders) | 1 (1)
bruising on forearms (Blood and lymphatic system disorders) | 1 (1)
chest pain (Musculoskeletal and connective tissue disorders) | 1 (1)
constipation (Gastrointestinal disorders) | 6 (6)
cough (Respiratory, thoracic and mediastinal disorders) | 5 (5)
creatinine (Blood and lymphatic system disorders) | 7 (7)
decreased appetite (Gastrointestinal disorders) | 5 (5)
decreased leukocytes (Blood and lymphatic system disorders) | 1 (1)
decreased performance status (General disorders) | 1 (1)
decreased renal perfusion (Renal and urinary disorders) | 1 (1)
dehydration (Gastrointestinal disorders) | 1 (1)
delirium (Nervous system disorders) | 1 (1)
depression (Psychiatric disorders) | 3 (3)
diarrhea (Gastrointestinal disorders) | 3 (3)
difficulty hearing (Ear and labyrinth disorders) | 1 (1)
dizziness (Nervous system disorders) | 5 (5)
dry eyes (Eye disorders) | 1 (1)
dry mouth (Gastrointestinal disorders) | 1 (1)
dry skin (Skin and subcutaneous tissue disorders) | 1 (1)
dysphagia (Gastrointestinal disorders) | 2 (2)
dyspnea (Respiratory, thoracic and mediastinal disorders) | 5 (5)
ear pain (Ear and labyrinth disorders) | 1 (1)
edema (Blood and lymphatic system disorders) | 5 (5)
elevated albumin (Blood and lymphatic system disorders) | 1 (1)
elevated ANC (Blood and lymphatic system disorders) | 1 (1)
elevated AST/ALT (Blood and lymphatic system disorders) | 1 (1)
fatigue (General disorders) | 14 (14)
febrile neutropenia (Infections and infestations) | 1 (1)
fever (Infections and infestations) | 4 (4)
gingivitis (General disorders) | 1 (1)
hyperglycemia (Endocrine disorders) | 14 (14)
granulcytopenia (Blood and lymphatic system disorders) | 1 (1)
headache (Nervous system disorders) | 2 (2)
heartburn (Gastrointestinal disorders) | 2 (2)
hydronephrosis (Renal and urinary disorders) | 1 (1)
hypernatremia (Blood and lymphatic system disorders) | 1 (1)
hypertension (Cardiac disorders) | 1 (1)
hypoalbuminemia (Gastrointestinal disorders) | 2 (2)
hypokalemia (Blood and lymphatic system disorders) | 4 (4)
hypocalcemia (Blood and lymphatic system disorders) | 1 (1)
hypomagnsmia (Blood and lymphatic system disorders) | 1 (1)
hypophosphatemia (Blood and lymphatic system disorders) | 1 (1)
hyponatremia (Blood and lymphatic system disorders) | 1 (1)
hypotension (Cardiac disorders) | 4 (4)
hypovolemia (Blood and lymphatic system disorders) | 1 (1)
infection (Infections and infestations) | 2 (2)
ingrown toenail (General disorders) | 1 (1)
chills (General disorders) | 1 (1)
itching (Skin and subcutaneous tissue disorders) | 2 (2)
joint pain (Musculoskeletal and connective tissue disorders) | 5 (5)
leukopenia (Blood and lymphatic system disorders) | 14 (14)
low albumin (Blood and lymphatic system disorders) | 2 (2)
low magnesium (Blood and lymphatic system disorders) | 2 (2)
low phosphorus (Blood and lymphatic system disorders) | 1 (1)
lymphopenia (Blood and lymphatic system disorders) | 1 (1)
malaise (General disorders) | 1 (1)
mucositis (Gastrointestinal disorders) | 1 (1)
nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 (2)
nausea (Gastrointestinal disorders) | 16 (16)
neuropathy (Nervous system disorders) | 1 (1)
neutropenia (Blood and lymphatic system disorders) | 28 (28)
night sweats (General disorders) | 2 (2)
dry cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
orthostatic hypotension (Cardiac disorders) | 1 (1)
palpitations (Cardiac disorders) | 1 (1)
paralytic ileus (Gastrointestinal disorders) | 1 (1)
pharyngitis (Gastrointestinal disorders) | 1 (1) — strep
protein calorie malnutrition (Metabolism and nutrition disorders) | 1 (1)
protein low (Metabolism and nutrition disorders) | 1 (1)
pruritis (Skin and subcutaneous tissue disorders) | 1 (1)
rash (Skin and subcutaneous tissue disorders) | 3 (3)
renal artery vasoconstruction (Renal and urinary disorders) | 1 (1)
right pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3 (3)
runny nose (Respiratory, thoracic and mediastinal disorders) | 2 (2)
SGOT (Blood and lymphatic system disorders) | 2 (2)
SGPT (Blood and lymphatic system disorders) | 4 (4)
shortness of breath (Respiratory, thoracic and mediastinal disorders) | 5 (5)
sinus problems (Respiratory, thoracic and mediastinal disorders) | 2 (2)
systoloc ejection murmur (Cardiac disorders) | 1 (1)
tachycardia (Cardiac disorders) | 3 (3)
bilirubin (Blood and lymphatic system disorders) | 2 (2)
thrombocytopenia (Blood and lymphatic system disorders) | 33 (33)
upper respiratory infection (Respiratory, thoracic and mediastinal disorders) | 2 (2)
vomiting (Gastrointestinal disorders) | 10 (10)
weakness (General disorders) | 5 (5)
weight gain (General disorders) | 1 (1)
weight loss (General disorders) | 1 (1)
wheezing (Respiratory, thoracic and mediastinal disorders) | 3 (3)
pain (General disorders) | 7 (7)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less